CLINICAL TRIAL: NCT04796818
Title: Evaluation of Treatment Response of Colorectal Cancer Liver Metastases With Intravoxel Incoherent Motion Diffusion Weighted Imaging
Brief Title: An Investigational Scan (Intravoxel Incoherent Motion Diffusion Weighted Imaging) for the Evaluation of Colorectal Cancer Liver Metastases Treatment Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0004; NCI-2020-07466 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0004 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-21; First posted 2021-03-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Carcinoma; Metastatic Malignant Neoplasm in the Liver; Resectable Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (IVIM DWI) (Experimental): Patients undergo IVIM DWI over 10 minutes during standard of care MRI within 30 days of starting chemotherapy and after 4-6 cycles of preoperative chemotherapy.
  Interventions: Procedure: Diffusion Weighted Imaging

INTERVENTIONS:
Procedure: Diffusion Weighted Imaging — Undergo IVIM DWI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DW-MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging

SUMMARY:
This trial evaluates the treatment response of colorectal cancer that has spread to the liver (liver metastases) using intravoxel incoherent motion diffusion weighted imaging (IVIM DWI). IVIM DWI is new kind of imaging scan that may help measure changes in disease before and after chemotherapy in patients with colorectal liver metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether intravoxel incoherent motion (IVIM) diffusion weighted imaging (DWI) can detect a difference between the changes in the diffusion related parameters in patients before and after chemotherapy between responders and nonresponders.

SECONDARY OBJECTIVES:

I. Use respiratory-triggered DWI and quantitative T2 maps for the evaluation of colorectal liver metastases (CLM) after treatment.

II. Assess whether changes in these parameters correlate to pathologic treatment response (percent necrosis) determined on pathology.

OUTLINE:

Patients undergo IVIM DWI over 10 minutes during standard of care MRI within 30 days of starting chemotherapy and after 4-6 cycles of preoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with treatment-naive resectable CLM, who will start chemotherapy with oxaliplatin with fluorouracil (5-FU)/leucovorin (FOLFOX), irinotecan with 5-FU/leucovorin (FOLFIRI), or a combination, such as fluorouracil, leucovorin, oxaliplatin and irinotecan (FOLFOXIRI), with or without a biologic agent
* Patients with at least 1 colorectal liver metastasis measuring at least 1 cm
* Patients with anticipated follow-up before and after surgery at MD Anderson

Exclusion Criteria:

* Patients who have already received preoperative chemotherapy for the CLM or will undergo radiation therapy, ablative therapies, or other non-surgical therapies directed at the liver
* Patients allergic to gadolinium
* Patients with pacemakers
* Greater than 400 pounds in weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change in the true diffusion coefficient (D) | Up to 3 months or 5 months (each cycle is 28 days)
  The absolute changes of parameter D between response and nonresponse groups will be compared using a two-sample t-test.

SECONDARY OUTCOMES:
Diffusion related parameters in intravoxel incoherent motion diffusion weighted imaging | Up to 3 months or 5 months (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Priya R Bhosale, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org